CLINICAL TRIAL: NCT04247360
Title: Effect of Cuff Pressure During Operation on Postoperative Sore Throat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Jiwon Lee, assistant professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-09-030
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cuff pressure with 20cmH2O (Other): continuous monitoring and maintaining cuff pressure with 20 cmH2O during surgery
  Interventions: Device: cuff pressure
- cuff pressure with 30cmH2O (Other): continuous monitoring and maintaining cuff pressure with 30 cmH2O during surgery
  Interventions: Device: cuff pressure

INTERVENTIONS:
Device: cuff pressure — maintaining cuff pressure according the groups

SUMMARY:
When general anesthesia is performed for surgery, tracheal intubation is performed. In order to ventilate after performing tracheal intubation, air is injected into the cuff attached to the tube to fill the gap between the tracheal tube and the patients's inner surface of trachea.

Even though, 20 to 30 cm H2O is known to be the appropriate pressure to prevent air leaks while preventing ischemic damage of tracheal mucosa. So, Researchers want to observe clinical differences in pressure at both ends of the safety zone of the cuff pressure.

DETAILED DESCRIPTION:
Patients who are scheduled for elective surgery/ general anesthesia are randomized to two groups.

l : cuff pressure - 20cmH2O ll : cuff pressure - 30cmH2O

After tracheal intubation with routine method, cuff pressure is continuously monitored with manometer. The anesthesia during surgery is maintained with 0.8 MAC of desflurane and continuous remifentanil. Clinical outcomes (sore throat, hoarseness and postoperative pain) are evaluated after 0 minutes, 2 hours, 4 hours, and 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing total hip replacement arthroplasty that require general anesthesia

Exclusion Criteria:

* a patient who disagrees with the study
* tracheal stenosis
* operation time > 3 hours or < 1 hour 30 minutes
* difficult airway
* drug abuse, alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
postoperative sore throat | At postoperative 24 hours
  Number of participants with postoperative sore throat for postoperative 24 hours

SECONDARY OUTCOMES:
postoperative hoarseness | At postoperative 24 hours
  Number of participants with postoperative hoarseness for postoperative 24 hours
nausea | At postoperative 24 hours
  Number of participants with postoperative nausea for postoperative 24 hours
Requirements of analgesics | At postoperative 24 hours
  Number of participants with analgesics use for postoperative 24 hours

IPD SHARING:
Plan to Share IPD: No